CLINICAL TRIAL: NCT01781845
Title: Evaluation of Ultrasound Acoustic Radiation Force Impulse (ARFI)Shear Wave Velocity Imaging (SVI)in the Characterization of Pediatric Hydronephrosis
Brief Title: Hydronephrosis ARFI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jonathan R. Dillman M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00064524
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Hydronephrosis
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARFI-SVI Ultrasound (Experimental): Ultrasound scan using acoustic radiation force impulse-shear wave velocity imaging in the characterization of pediatric hydronephrosis. This is a non-invasive scan that uses sound waves to create the images.
  Interventions: Procedure: AFRI-SVI Ultrasound

INTERVENTIONS:
Procedure: AFRI-SVI Ultrasound — This research scan uses acoustic radiation force impulse (ARFI) shear wave velocity imaging (SVI)a new ultrasound technology in which unique sound waves create the images/pictures of the kidney beng examined/scanned. This ultrasound scan will take approximately 10 minutes to complete.

SUMMARY:
Pediatric upper urinary tract dilatation (hydronephrosis) is relatively common and may be either obstructive or nonobstructive. While the upper urinary tract is commonly evaluated by ultrasound, this imaging technique often fails to distinguish obstructed from nonobstructed systems. ARFI SVI is a new ultrasound technology that can be used to determine stiffness by measuring a tissue's shear wave velocity, may show alterations in parenchymal shear wave velocity in kidneys that show obstruction on DRS (Diuretic renal scintigraphy)which serves as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or younger
2. You are scheduled for diuretic scintigraphy (DRS)testing -

Exclusion Criteria:

None

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
ARFI-SVI | 6 months
  fibrosis and intratubular pressure will be evidenced by higher parenchymal shear wave velocity measurements using the ARFI-SVI technology.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States